CLINICAL TRIAL: NCT02108691
Title: Effect of Intake of Glycin Max (L.) Merr. Peel Extract on Body Fat and Body Weight
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yongsoon Park, Associate Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SSWU-BF-GE
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycin max(L.) Merr. pell extract (Experimental)
  Interventions: Dietary Supplement: Glycin max(L.) Merr. peel extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Glycin max(L.) Merr. peel extract — Glycin max(L.) Merr. peel extract (2.5g/day)
  Arms: Glycin max(L.) Merr. pell extract
Dietary Supplement: Placebo — Placebo (2.5g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 8-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Glycin max (L.) Merr. peel extract on decrement of body fat. The investigators measured decrement of body fat parameters , including Body Fat Mass, Percent Body Fat, weight and BMI(body mass index), and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-65 years old
* BMI(body mass index) ≥ 25 kg/m^2 or WC(Waist Circumference) ≥ 90(men), WC ≥ 85(women)
* Able to give informed consent

Exclusion Criteria:

* Significant variation in weight(more 10%) in the past 3 months
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Started | 40 | 40
Completed | 32 | 31
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.30 (9.42) | 30.88 (9.18) | 30.59 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Fat Mass
Description: Body Fat Mass was measured in study visit 1(0 week) and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
g
  0 week | 16790.27 (3524.04) | 18223.75 (5325.29)
  8 week | 20174.10 (4336.18) | 21474.88 (6042.38)

2. Secondary Outcome: Changes in Percent Body Fat
Description: Percent Body Fat was measured in study visit 1(0 week) and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
percentage
  0 week | 24.28 (6.44) | 25.15 (7.92)
  8 week | 28.52 (7.44) | 28.76 (8.58)

3. Secondary Outcome: Changes in Weight
Description: Weight was measured in study visit 1(0 week)and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
kg
  0 week | 78.50 (10.89) | 81.46 (9.59)
  8 week | 77.36 (10.89) | 80.60 (9.57)

4. Secondary Outcome: Changes in BMI(Body Mass Index)
Description: BMI(body mass index) was measured in study visit 1(0week) and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
kg/m^2
  0 week | 27.62 (1.63) | 28.29 (1.91)
  8 week | 27.22 (1.77) | 28.00 (2.04)

5. Secondary Outcome: Changes in LDLc
Description: LDLc was measured in study visit 1(0week) and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
mg/dl
  0 week | 122.50 (33.71) | 113.81 (35.16)
  8 week | 98.47 (23.91) | 104.06 (24.39)

6. Secondary Outcome: Changes in Non-HDLc
Description: Non-HDLc was measured in study visit 1(0week) and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
mg/dl
  0 week | 171.63 (38.08) | 166.52 (46.45)
  8 week | 128.78 (32.19) | 137.39 (37.24)

7. Secondary Outcome: Changes in LDLc/HDLc
Description: LDLc/HDLc was measured in study visit 1(0week) and visit 3(8 week).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Number analyzed (Participants) | 32 | 31
ratio
  0 week | 2.21 (0.64) | 2.04 (0.57)
  8 week | 2.02 (0.60) | 2.15 (0.58)

ADVERSE EVENTS:
Arm/Group | Glycin Max(L.) Merr. Pell Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes